CLINICAL TRIAL: NCT05930119
Title: A Phase 1, Open-label, 4-period, Randomized 6-sequence Study to Evaluate the Effect of Food and Rabeprazole, a Proton Pump Inhibitor, on the Pharmacokinetics of HMPL-453 in Healthy Volunteers
Brief Title: HMPL-453 Food Effect and PPI Study in Healthy Volunteer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-453-00CH1
Record Dates: First submitted 2023-05-22; First posted 2023-07-05 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Rabeprazole

STUDY DESIGN:
Intervention Model Description: Open-label, 4-Period, Randomized 6-Sequence Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- fast overnight (Experimental): Subjects in treatment A will administered HMPL-453 at fast overnight condition.
  Interventions: Drug: HMPL-453
- high-fat meal (Experimental): Subjects in treatment B will administered HMPL-453 at high-fat meal condition.
  Interventions: Drug: HMPL-453
- low-fat meal (Experimental): Subjects in treatment C will administered HMPL-453 at low-fat meal condition.
  Interventions: Drug: HMPL-453
- rabeprazole (Experimental): Subjects in treatment D will administered rabeprazole combined with HMPL-453 at low-fat meal condition hour prior to receiving a standardized low-fat meal.
  Interventions: Drug: HMPL-453; Drug: Rabeprazole

INTERVENTIONS:
Drug: HMPL-453 — 300 mg HMPL-453
Drug: Rabeprazole — 20 mg of rabeprazole will be administered by mouth once daily.
  Arms: rabeprazole

SUMMARY:
A Phase 1, Open-label, 4-Period, Randomized 6-Sequence Study to Evaluate the Effect of Food and Rabeprazole, a Proton Pump Inhibitor, on the Pharmacokinetics of HMPL-453 in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent form;
2. The volunteer is male or female between the ages of 18 and 55 years old (inclusive) at the time of informed consent.
3. The volunteer has a body mass index (BMI)>18 and ≤29.9 kg/m2at screening. Male need≥50 kg，famele need≥45 kg.
4. Female with fertility agree to adopt efficient contraceptive measures within 6 months after signing ICF until the end of the last HMPL-453 dosing, and agree not to donate eggs (or oocytes) for reproductive purposes during this period. Acceptable and efficient contraceptive methods include complete abstinence, bilateral tubal ligation, oral or injection contraceptives, intrauterine devices, or partner vas deferens ligation. All hormonal contraception measures must be combined with barrier measures such as the use of condoms by spouses. More information can be found in Attachment 12.3 [Definition of Women with Fertility (WOCBP) and Acceptable and Unacceptable Contraceptive Methods].
5. Male patients is willing to take contraception measures (during the study and for 3 months after the end of study treatment). Male patients should avoid donating or freezing sperm during this period.
6. The volunteer is willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. The volunteer has a known history of any gastrointestinal surgery or any condition possibly affecting drug absorption (eg, cholecystectomy, gastrectomy, achlorhydria, peptic ulcer disease, or history of stomach or intestinal surgery or resection).
2. The volunteer had a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
3. The volunteer has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or at Day -1 check-in (baseline).
4. The volunteer has systolic blood pressure >140 mmHg diastolic blood pressure >90mmHg.
5. Currently keratopathy confirmed by ophthalmological examination, including but not limited to bullae keratopathy, zonal corneal degenerations, corneal abrasion, corneal ulcer, and sclerokeratitis.
6. Current or prior history of retinal detachment.
7. The volunteer has a clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval >480msec), or hasa family history of prolonged QTc syndrome or sudden death.
8. Volunteers who smoke more than 10 cigarettes per day within the first 3 months of screening and are unable to completely quit smoking during the study period.
9. Volunteers who frequently drink alcohol within the first 6 months before screening, drink more than 14 units of alcohol per week。
10. The volunteer has a history of drug misuse within 6 months prior to screening (including those who have tested positive for morphine, methylenedioxymethamphetamine, methamphetamine, tetrahydrocannabinol acid, ketamine, cocaine, or a positive urine drug test at screening or at check-in).
11. The volunteer has been diagnosed with acquired immune deficiency syndrome or has performed tests that are positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
12. The volunteer has a clinically significant X-ray,
13. The volunteer has participated in a clinical trial of other study drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the volunteer is currently enrolled in another clinical trial.
14. The volunteer has used CYP3A strong inducer or strong inhibitor, any over-the-counter (OTC) medications or prescription drugs (medications that can lower gastric acid in particular) within 2 weeks prior to the first dose.
15. The volunteer has consumed alcohol, grapefruit, lime, and caffeine within 72 hours prior to the first dose.
16. Taking drugs or dietary supplements (such as calcium, phosphorus, vitamin D, parathyroid hormone, etc.) that may cause blood phosphorus and/or blood calcium to rise within 2 weeks prior to the start of the study treatment.

18.Needle sickness, blood sickness or difficulty in collecting venous blood. 19.The volunteer is allergic to any of the study drugs (or its excipients) to be given in this study.

20.A female participant is pregnant, lactating, or breastfeeding. 21.Any other medical condition judged by the investigator would make the patients unsuitable to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
PK parameter for HMPL-453: AUC0-t | Day 1 to Day 33
  Area under the concentration time curve from time 0 to the last measurable concentration
PK parameter for HMPL-453: AUC0-inf | Day 1 to Day 33
  Area under the concentration time curve from time 0 extrapolated to infinity
PK parameter for HMPL-453: Cmax | Day 1 to Day 33
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Assessment of safety procedures findings | Day 1 to Day 33
  Any untoward medical occurrence associated with the study drug
PK parameter for HMPL-453: tmax,t1/2 | Day 1 to Day 33
  Time to reach the maximum observed plasma concentration, elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China